CLINICAL TRIAL: NCT01036516
Title: PET Assays of Striatal Dopamine Markers in Cocaine Craving
Brief Title: PET Assays of Striatal Dopamine Marker in Cocaine Craving
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998391; 98-DA-N391
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-27

CONDITIONS: Neural Systems; Drug Abuse; Cocaine Dependence
Keywords: Drug Cues; Dopamine Release; Psychomotor Stimulants; D2 Dopamine Receptor Subtype; Neuroimaging
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Cues related to past drug use induce a particular pattern of brain activation, which has been correlated with craving for cocaine in active cocaine abusers. Researchers are interested in determining the role of the brain chemical dopamine in cue-elicited as well as spontaneous craving for cocaine.
* To study the role of dopamine in cocaine craving, researchers will use positron emission tomography (PET) to compare the neural reactions of cocaine users with those of non-substance-abusing healthy volunteers. Researchers hope that the data gathered from this study will lead to the development of more effective anti-craving medications.

Objectives:

* To clarify the role of dopamine in cue-elicited responses that contribute to cocaine abuse.
* To determine if PET results of this study differ with various means of administering PET chemicals.

Eligibility:

- Individuals 21 to 44 years of age who are either current cocaine users (at least twice per week) or healthy volunteers without a history of drug abuse.

Design:

* Cocaine-using participants will enter the inpatient clinical research ward at the National Institute on Drug Abuse (NIDA) Addiction Research Center for 2 nights before the day of the study. In addition, these participants will stay overnight at NIDA the evening after each PET session and will be discharged the following day. Cocaine-using participants will be required to perform a balance test before the study to provide a baseline response in case they require anti-anxiety medications to cope with the effects of the study.
* Control subjects will not be required to stay overnight and will arrive as outpatients for the PET session. All participants will be required to abstain from alcohol and caffeine consumption from midnight before each study session, and will not be permitted to smoke on the day of testing.
* - On the day of the study, participants will undergo a practice session to set up the PET scanning equipment. Following the practice session, participants will be shown video recordings of images that are related to nature (e.g., seashells) or to drug abuse (e.g., drug paraphernalia). Participant reactions will be studied through the PET monitoring, and the study will be conducted in two separate PET sessions with a break in between. Individuals in the cocaine-using group may receive anti-anxiety medication if the stimulus cues increase anxiety related to cocaine craving.
* Different groups of participants will receive different methods of PET chemical administration, and researchers will compare these methods.

DETAILED DESCRIPTION:
Cues related to past drug use induce a particular pattern of brain activation, which has been correlated with craving for cocaine in active cocaine abusers. The proposed research is designed to assess the role of dopamine in cue-elicited as well as spontaneous craving for cocaine. Cocaine abusers and control subjects will be presented with a stimulus complex related to drug abuse (cocaine cues: videotape depicting drug use, drug paraphernalia) or to nature (neutral cues: videotape depicting items such as shells and pinecones). The effects of each cue condition on striatal D2-like dopamine (DA) receptors and changes in intrasynaptic dopamine will be measured by positron emission tomography (PET). The PET data will then be correlated with subjective self-reports of mood, particularly measures of craving. These results will be compared between the two subject groups. This research will help clarify the role of dopamine in cue-elicited responses that contribute to cocaine abuse. Ultimately, the results obtained may lead to the development of anti-craving medications.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: Subjects in both the cocaine abuser and control groups will be volunteers of either gender, aged 21 to 44 years.
  2. History of Drug Abuse: For the cocaine abuser group, regular current use of cocaine is required (at least twice per week) that has been ongoing for at least two years.

EXCLUSION CRITERIA:

1. Psychiatric disease: DSM IV criteria will be used. No subject with a current axis I diagnosis other than a substance abuse disorder will be allowed. No subject with a lifetime history of a schizophrenic disorder will be allowed.
2. History of Drug Abuse: Cocaine users will be excluded if toxicology screen at the time of obtaining informed consent is positive for any illicit drug other than cocaine. Volunteers for the control group with any history of intravenous drug abuse or any history of psychostimulant drug abuse will be excluded. Axis I diagnoses of substance abuse disorders other than nicotine abuse and/or dependence will be exclusionary criteria for volunteers in control group.
3. CNS disease: Structural brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), history of other neurological disease, or history of head trauma (defined as loss of consciousness > 2 min or requiring hospitalization).
4. Cardiovascular disease: Advanced coronary artery disease, endocarditis or other cardiac disease likely to result in cerebral embolism.
5. Pulmonary disease: Significant obstructive pulmonary disease, tuberculosis, or bronchospasm (asthma, emphysema, bronchitis).
6. Systemic disease: Endocrinopathies, renal or hepatic failure, or autoimmune disease involving the CNS.
7. Miscellaneous: Hematocrit < 35-36 (for women) or < 39 (for men), prostatic hypertrophy or chronic inflammation.
8. Claustrophobia: Subjects will be questioned about their potential discomfort in being in an enclosed space, such as a PET or MRI scanner.
9. Because of the potentially harmful effects of radiation exposure to fetuses and infants, female subjects who are pregnant, nursing, planning to become pregnant or who do not show evidence of reliable birth control will be excluded from participation.
10. Arterial circulation to the hand: Evidence of inadequate patency of radial and ulnar arteries, determined by either Doppler flow measurements or a positive Allen's test, is an exclusionary criterion for insertion of an arterial catheter. Potential subjects who do not have adequate arterial circulation in their hand but otherwise meet criteria could be included in this study and have only venous blood samples drawn.
11. Radiation exposure: Any subject who has had sufficient prior radiation exposure for research purposes (i.e., apart from medical procedures for diagnostic or therapeutic purposes) prior to beginning the study that exceeds 5.0 rem during the previous 12 months or 3.0 rem during the previous 3 months will be excluded.
12. Other medication: Volunteers who are currently taking any psychoactive medication, or are currently prescribed other drugs that affect central neurotransmitter systems, will be excluded from this study.
13. HIV positive individuals will be excluded because HIV infection and the development of AIDS produces abnormalities in brain function, and in particular in the basal ganglia (Rottenberg et al., 1987), where we propose to make measurements of [11C] raclopride binding.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 1998-06-23; Study Completion 2012-03-27

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Collins, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Berger SP, Hall S, Mickalian JD, Reid MS, Crawford CA, Delucchi K, Carr K, Hall S. Haloperidol antagonism of cue-elicited cocaine craving. Lancet. 1996 Feb 24;347(9000):504-8. doi: 10.1016/s0140-6736(96)91139-3. PMID 8596268
- [Background] Breier A, Su TP, Saunders R, Carson RE, Kolachana BS, de Bartolomeis A, Weinberger DR, Weisenfeld N, Malhotra AK, Eckelman WC, Pickar D. Schizophrenia is associated with elevated amphetamine-induced synaptic dopamine concentrations: evidence from a novel positron emission tomography method. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2569-74. doi: 10.1073/pnas.94.6.2569. PMID 9122236